CLINICAL TRIAL: NCT02526121
Title: Effect of Therapeutic Phlebotomies on the Triglycerides Concentration in Patients With Hypertriglyceridemia and Hyperferritinemia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Aragones de Ciencias de la Salud (Other Government)
Responsible Party: Principal Investigator, Fernando Civeira, Professor, Instituto Aragones de Ciencias de la Salud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEICA;PI10/099
Record Dates: First submitted 2015-03-25; First posted 2015-08-18 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Hyperferritinemia; Hypertriglyceridemia
MeSH Terms: conditions — Hyperferritinemia; Hypertriglyceridemia | interventions — Phlebotomy; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phlebotomy associated with dietary and lifestyle counseling (Experimental)
  Interventions: Procedure: Phlebotomy; Behavioral: Dietary and lifestyle counseling.
- Dietary and lifestyle counseling. (Active Comparator)
  Interventions: Behavioral: Dietary and lifestyle counseling.

INTERVENTIONS:
Procedure: Phlebotomy — Volume of 400 mL every 3 weeks, 3 times.
  Arms: Phlebotomy associated with dietary and lifestyle counseling
Behavioral: Dietary and lifestyle counseling. — Dietary and lifestyle counseling.

SUMMARY:
The purpose of this study is to evaluate the effect of iron depletion with phlebotomies on blood triglyceride concentration, in subjects with hypertriglyceridemia and iron overload, compared with a dietary intervention alone.

All subjects in this study will follow dietary and lifestyle counseling in a period of 3 months.

A randomized group will receive phlebotomies every 3 weeks in this period.

ELIGIBILITY:
Inclusion Criteria:

* Hyperferritinemia: > 300µgr/L for male and >200µgr/L for female.
* Hypertriglyceridemia: > 200 mg/dL in two determinations after at least ten hours of fasting and lipid-lowering diet.

Exclusion Criteria:

* Contraindications for phlebotomy: poor venous access, previous intolerance (hypotension or apprehension), heart disease, anemia.
* Subjects suffering from acute or chronic disease, including liver disease, diabetes, cancer, kidney disease or uncontrolled thyroid disease.
* Elevated C reactive protein (CRP) as a parameter of inflammation (>10mg/L).
* Alcohol intake: over 30 gr. per day for men and 25 gr. per day for women.
* Lipid lowering drugs use.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Triglycerides concentration | Three months before

SECONDARY OUTCOMES:
Iron parameters | Three months before
  Ferritin level: >300 µgr/L in men and >200 µgr/L in women

OTHER OUTCOMES:
Total cholesterol | Three months before
HDL-cholesterol | Three months before
LDL- cholesterol | Three months before
Apolipoprotein A1 | Three months before
Apolipoprotein B | Three months before
Peripheral Insulin resistance measured by HOMA | Three months before
Inflammatory cytokines | Three months before
C Reactive Protein | Three months before

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Civeira, MD, PhD, Principal Investigator — Unidad de Lípidos/ Laboratorio de Investigación Molecular; Hospital Universitario Miguel Servet; Instituto Aragonés de Ciencias de la Salud (Zaragoza, Spain)
Locations (1):
- Hospital Universitario Miguel Servet, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Mateo-Gallego R, Lacalle L, Perez-Calahorra S, Marco-Benedi V, Recasens V, Padron N, Lamiquiz-Moneo I, Baila-Rueda L, Jarauta E, Calmarza P, Cenarro A, Civeira F. Efficacy of repeated phlebotomies in hypertriglyceridemia and iron overload: A prospective, randomized, controlled trial. J Clin Lipidol. 2018 Sep-Oct;12(5):1190-1198. doi: 10.1016/j.jacl.2018.06.017. Epub 2018 Jul 4. PMID 30049591